CLINICAL TRIAL: NCT04047485
Title: Evaluation of the Effect of Cataract Surgery on Cognitive Function in Very Elderly Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Gian Maria Cavallini, Associate Professor, Head of Ophthalmology, Director, School of Specialization in Ophthalmology., University of Modena and Reggio Emilia
Other Study IDs: 1005/2018/OSS/AOUMO
Record Dates: First submitted 2019-07-25; First posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Dementia; Mild Cognitive Impairment; Cataract Senile; Cataract; Delirium in Old Age; Delirium Confusional State; Post-Op Complication; Cataract in Old Age
Keywords: Cataract; Mild Cognitive Impairment (MCI); Cataract Surgery; BMICS (Bi-Manual Microincisional Cataract Surgery); Post-operative Delirium
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Cataract; Confusion; Postoperative Complications; Emergence Delirium | interventions — Visual Acuity; Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Elderly Female (A): Female subjects between 65 and 85 years old
  Interventions: Diagnostic Test: Visual Acuity; Diagnostic Test: CAM (Confusion Assesment Method); Diagnostic Test: CATQUEST 9-SF; Diagnostic Test: OCT; Diagnostic Test: 6CIT; Diagnostic Test: Barthel Index; Diagnostic Test: Endothelial Microscopy - Cornea
- Great Elderly Female (B): Female subjects with more than 85 years old
  Interventions: Diagnostic Test: Visual Acuity; Diagnostic Test: CAM (Confusion Assesment Method); Diagnostic Test: CATQUEST 9-SF; Diagnostic Test: OCT; Diagnostic Test: 6CIT; Diagnostic Test: Barthel Index; Diagnostic Test: Endothelial Microscopy - Cornea
- Elderly Male (C): Male subjects between 65 and 81 years old
  Interventions: Diagnostic Test: Visual Acuity; Diagnostic Test: CAM (Confusion Assesment Method); Diagnostic Test: CATQUEST 9-SF; Diagnostic Test: OCT; Diagnostic Test: 6CIT; Diagnostic Test: Barthel Index; Diagnostic Test: Endothelial Microscopy - Cornea
- Great Elderly Male (D): Men subjects with more than 81 years old
  Interventions: Diagnostic Test: Visual Acuity; Diagnostic Test: CAM (Confusion Assesment Method); Diagnostic Test: CATQUEST 9-SF; Diagnostic Test: OCT; Diagnostic Test: 6CIT; Diagnostic Test: Barthel Index; Diagnostic Test: Endothelial Microscopy - Cornea

INTERVENTIONS:
Diagnostic Test: Visual Acuity — During T0, T2 and T3, every subject has been evaluated with a Snellen Chart, to measure visual acuity in number of letters (BVCA)
Diagnostic Test: CAM (Confusion Assesment Method) — During the first 48 hours of post-op follow-up, any episode of "post-operative Delirium" is checked and evaluated.
Diagnostic Test: CATQUEST 9-SF — The questionnaire contains questions evaluating the benefits of cataract surgery. The questionnaire has been used during T0, T2 and T3
Diagnostic Test: OCT — Using the RNFL and the Macular Topography protocol, the macula and optical nerve are measured during the T2 phase of each patient the risk of Irvine Gas's syndrome or any other retinal complication.
  Other Names: Optical Coherence Tomography
Diagnostic Test: 6CIT — This Cognitive Impairment test doesn't require Visual function to be executed. Cognitive function is evaluated at T0, T1 and the post-operative trend at T2 and T3.
  Other Names: Kingship Test
Diagnostic Test: Barthel Index — To evaluate the everyday independence of the subject and it's trend durin the follow-up
Diagnostic Test: Endothelial Microscopy - Cornea — Endothelial cell density is evaluated before surgery (T0) and during the follow-up (T2 and T3). The reason of the choice of this test is to evaluate the trend of these instrumental parameters in the elderly population.

SUMMARY:
The study intends to measure the evolution over time of the cognitive capacity of patients undergoing cataract surgery in relation to the opaque lens removal surgery (cataract) in a population considered to be at risk of neurocognitive degeneration.

Secondary objectives:

• Estimate the incidence of postoperative cognitive dysfunctions and any episodes of perioperative delirium with the aim of demonstrating the safety of cataract surgery in the elderly patient in terms of cognitive functions and impact on the psychological state.

In the context of the study a risk sub-population analysis will be carried out, evaluating the trend over time of the "endothelial cells count" parameter

The elderly population remains, due to the aging of the cornea, a population "at risk" for significant alterations from the clinical point of view. During the study the endothelial cells count will be monitored, in order to be able to evaluate the safety of the cataract surgery and to be able to correctly correlate a possible deterioration in the visual acuity of patients with corneal decompensation. To evaluate the progress of the endothelial cells count in the elderly patient during the pre-intervention and post-intervention period. Since the low values of cellular media in endothelial microscopy are an element that increases the risk of complications during cataract surgery, the study wants to assess how waiting times between filter visits and cataract surgery can cause an elderly patient worsening of this parameter even in a few months. The trend of the same parameter will be monitored even after the intervention since in case of decrease, the low endothelial count could cause an alteration of visual acuity and therefore a minor improvement in cognitive performance.

The research will be set as a longitudinal observational study where will be compared in each patient the parameters analyzed in the 6 months prior to cataract surgery and in the 3 months following the operation itself. Patients will be enrolled during the first cataract filter visit, will be submitted to simple questions and their clinical data will be collected. Subsequently, before and after three months of surgery repeated cognitive testing and the control normally performed instrumental tests during follow-up.

A clinical follow-up will be provided, during normal follow-up visits at 20 days and 6 months after the patient's surgery: the following information will be collected during these visits

* BCVA (visual acuity)
* endothelial cells microscopy
* OCT macula and optic nerve
* Catquest 9SF;
* Barthel Index;
* Six Item Cognitive Test
* Confusion Assessment Method (CAM): this exam will be performed within 24 hours of post-surgery and 20 days after surgery.

It is important to underline that the cognitive tests proposed to patients consist of simple questions that do not depend on the visual ability of the subject.

DETAILED DESCRIPTION:
Study design: prospective, monocentric, epidemiological study: non-interventional. The drafting of the protocol follows the order proposed by the STROBE check-list for the publication of the observational studies where applicable.

There is no agreement between promoter and clinical center.

There is no agreement between promoter and financier: the study has no funding. The study is also carried out for the purpose of completing a thesis.

Rational

The constant aging of the population in western countries has led to an increase in the incidence of visual deficits in the elderly, the incidence of cataract is around 68%, at the same time this category of subjects frequently has cognitive deficits that can be minimal or severe as in the case of dementias.

The individual's visual capacity is correlated with the neurological progression of these morbid states. Numerous studies have long sought a correlation between sensory (visual and auditory) functionality and cognitive faculties in old age, defining how sensory functions can be considered indicators of the integrity of the central nervous system.

Further studies, always focused on this current research, focused on a correlation between the improvement of visual acuity through the IOL (Intra Ocular Lens) implant and the improvement of cognitive faculties. Further studies have focused their attention not only on cognitive faculties, but on the psychological aspect in terms of improving the quality of life following cataract surgery. Simultaneously, Cataract surgery has been referred as one the most effective healthcare intervention to prevent and lower the risk of falls, hips and lower limbs fracture, trauma and social isolation.

The improvement of the visual capacity, the cognitive faculties and the psychological state of the elderly patient are certainly useful elements for improving the quality of life of the subject but also for the caregiving burden on the elderly patient by the caregivers and the NHS. A 1998 study found a strong association between visual impairment (caused by altered contrast sensitivity, reduced field of vision and the presence of cataracts) and the increase in falls in the elderly.

Materials and methods

Patients will be enrolled during the filter visits of the ophthalmology clinic: whenever the need for replacement of the operative lens will be diagnosed, the patient will be offered to participate in the data collection by providing the information sheet. Subsequently consent will be collected. Data collection will be undertaken when the consent is signed. An identification code will be assigned exclusively to each patient. The patient's personal data will be entered through the creation of the Patient's list, to keep personal data confidential.

In no case will experimental treatments be provided to the patient: the study includes a collection of clinical information already normally collected during preoperative visits, outpatient visits and during follow-up checks.

The research will be set as a longitudinal observational study where will be compared in each patient the parameters analyzed in the 6 months prior to the cataract operation and in the 3 months following the operation itself.

The cognitive state will be measured over time: during enrollment, on the day of surgery, 20 days after surgery and 3 months after surgery.

Patients will be enrolled during the first cataract filter visit, will be submitted to simple questions and their clinical data will be collected.

A comparison will also be made in terms of incidence of neuro-cognitive and delirium problems in relation to the patient's age and cataract surgery. The great elderly population has a higher risk to encounter a momentaneous cognitive disfunction, due to psycological and physical stress induced by surgery and anesthesia. This study, considering this important element, will indirectly estimate the safety of cataract surgery. The post-operative delirium incidence in a surgical ward is considered an important parameter of quality of care in terms of patient's care and technical management in the ward.

The information sheet will be provided during the filter visit for the insertion of the patient on the waiting list for cataract surgery and consent will be collected after this.

The following parameters will be analyzed: demographic variables, level of education, presence of relatives during the visit, patient history of proximal and remote patient, home therapies, performed analyzes of practice during outpatient visits: BCVA visual acuity (ETDRS optotype tables), microscopy endothelial, OCT macula and optic nerve to exclude the presence of a maculopathy and a deficit of nerve fibers such as to affect the improvement of visual and cognitive function.

Following the collection of the consent, questionnaires will be provided to the patients enrolled to measure the functional cognitive capacity of the subject such as:

Quality of life, Catquest 9SF. The Catquest evaluation consists of 9 questions, evaluating the perceived quality of vision in routine activities like reading, shopping, recognizing individuals or doing recreational activities. The 9 questions present a speicific scale of 5 measures, from "Great Difficult" to "No difficult". The rationale beneath this test is to evaluate the ratio between the personal perception of visual function before and after surgery, evaluating in parallel trends of the mean of the scores calculated. A comparison will be also set between eleders and great elders, to evaluate eventual differences between the perceived result of surgery and the real visual acuity.

Scale of evaluation of daily life activity, Barthel Index. Many clinical studies associated the surgical removal of opacified lens with an increase of independence, due to the increase of visual function. To measure eventual changes, the Barthel Index has been chosen and added inside the protocol. The Barthel scale is an ordinal scale used to measure performance in activities of daily living (ADL). Each performance item is rated on this scale with a given number of points assigned to each level or ranking. This test is used by general physicians, physiotherapists, neurologists and rehabilitation nurses to calculate the trend of physical independence of an individual. This Index evaluates the physical necessities in daily activities like personal hygiene, Mobility, feeding, dressing, bladder control and bowels. The evaluation in this case consists on a score between 0-100 where 100 means complete independence and 0 absolute dependence on someone else.

Cognitive state measured with the Six Item Cognitive Impairment Test (6CIT). Number of questions: 6. Time taken to perform: 3-4 minutes. Score: the 6CIT uses an inverse score and questions are weighted to produce a total out of 28. Scores of 0-7 are considered normal and 8 or more significant. Advantages: the test has high sensitivity without compromising specificity, even in mild dementia. It is easy to translate linguistically and culturally. Disadvantages: the main disadvantage is in the scoring and weighting of the test, which is initially confusing; however, computer models have simplified this greatly.

Probability statistics: at the 7/8 cut-off: Overall figures - sensitivity = 90%, specificity = 100%; in mild dementia, sensitivity = 78%, specificity = 100%. Differently from older studies, the choice of this evaluation method The quickness of the administration of the test and more importantly, the exclusive use of question, and not the use of visual function provides to the study a more complete and purified view of the cognitive function, configuring this study as a innovation in the field.

Following the secondary outcomes, the corneal behavior will be measured between the different groups, focusing on the age criteria. Considering a physiological lowering of the quality of the cornea, the phacoemulsification is a physical stress for the ocular structure, raising the risk of corneal decompensation. To tangibly measure the corneal behavior, corneal thickness and corneal endothelial cells density have been chosen as main parameters. The CSO Perseus 400 (Florence - IT) will be used to study corneal behavior.

At the same time, the Optical Coherence Tomography will be used to evaluate the Macula and the optical nerve modifications after cataract surgery. This evaluation will be set in the highest risk period (up to 30 days after cataract surgery). The Irvine Gass macular edema and optical nerve insults can be a cause of lower visual improvement after a correct cataract surgery. The OPKO OCT/SLO will be used to conduct these measures.

Study Phases and Times

Time 0: patient enrollment (on average 4 months before surgery) Time 1: perioperative time Time 2: check at 20 days Time 3: check at 3 months

It is important to underline that the cognitive tests proposed to patients consist of simple questions that do not depend on the visual ability of the subject.

Finally, the study will compare the incidence data of neuro-cognitive problems in those who have undergone surgery in relation to the patient's age group and cataract surgery.

Data are analyzed using the R-Software, and using the ANOVA calculation method. Analysis of variance (ANOVA) is a collection of statistical models and their associated estimation procedures (such as the "variation" among and between groups) used to analyze the differences among group means in a sample. With this analysis, the trend of each variable will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age ≥ 65 years undergoing cataract surgery. Cataract surgery is indicated by the medical-scientific community according to good clinical practice and not influenced by the study's criteria. The purpose of the study is to add clinical-scientific information of any relevance.

Exclusion Criteria:

* Patient refusal
* Diagnosis of dementia by the specialist in neurocognitive diseases (neurologist and / or geriatrician)
* maculopaties and other ophthalmopaties (according to diagnosis of ophthalmologist specialist) because the visual capacity is invalidated regardless of the opacification of the crystalline and therefore the cognitive function is not affected by a post-intervention improvement.
* Patients who have performed cataract surgery in at least one eye since the previous cataract operation may have already caused changes in cognitive function causing confusion about the results of the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The studied population consists in people who can really obtain a visual acuity recovery with cataract surgery. All the variables are measured in a very elderly population (high risk population) and compared them in a elderly population (lower risk)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-02 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between visual acuity and cognitive function at 3 months after Cataract Surgery. | 6 months before surgery to 3 months after surgey
  The visual acuity trend and the cognitive function using the Kingshill (6CIT) score are measured during every visit. The 6 Item Cognitive Impairment Test (6CIT) is a test that doesn't provide the visual function. The choice of this kind of test resides in the capability of evaluating the cognitive function without any influence caused by cataract. The score is composed by 6 questions which evaluate the work memory, the temporal and spatial orientation. The test's result is a score, with a clinical cut-off of 7 points. The more points the subject makes, the higher risk of cognitive impairment is configured.
  The visual acuity is calculated with Snellen Chart using the Best Corrected Visual Acuity (BCVA) with the number of letters read.

SECONDARY OUTCOMES:
Post operative delirium prevalence | Only during the perioperative period (day of cataract surgery and the next 48 hours)
  The prevalence of post operative delirium is measured using the Confusion Assessment Method Evaluation.
Corneal endothelial cells density | 6 months before surgery, 20 days after cataract surgery and 3 months after cataract surgery.
  Thanks to the Endothelial Microscopy Evaluation, the corneal performance will be measured in terms of density of endothelial cells
Corneal pachymetry | 6 months before surgery, 20 days after cataract surgery and 3 months after cataract surgery.
  Thanks to the Corneal Pachymetry, the corneal performance will be measured in terms of density of corneal thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Gian Maria Cavallini, Associate Professor, Principal Investigator — Dipartimento Chirurgico, Medico, Odontoiatrico e di Scienze Morfologiche con interesse Trapiantologico, Oncologico e di Medicina Rigenerativa - UNIMORE - University of Modena and Reggio Emilia
Locations (1):
- Policlinico di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferri CP, Prince M, Brayne C, Brodaty H, Fratiglioni L, Ganguli M, Hall K, Hasegawa K, Hendrie H, Huang Y, Jorm A, Mathers C, Menezes PR, Rimmer E, Scazufca M; Alzheimer's Disease International. Global prevalence of dementia: a Delphi consensus study. Lancet. 2005 Dec 17;366(9503):2112-7. doi: 10.1016/S0140-6736(05)67889-0. PMID 16360788
- [Background] Jefferis JM, Mosimann UP, Clarke MP. Cataract and cognitive impairment: a review of the literature. Br J Ophthalmol. 2011 Jan;95(1):17-23. doi: 10.1136/bjo.2009.165902. Epub 2010 Aug 31. PMID 20807709
- [Background] Brookmeyer R, Johnson E, Ziegler-Graham K, Arrighi HM. Forecasting the global burden of Alzheimer's disease. Alzheimers Dement. 2007 Jul;3(3):186-91. doi: 10.1016/j.jalz.2007.04.381. PMID 19595937
- [Background] Taiel-Sartral M, Nounou P, Rea C, el Alamy A, Bendeddouche K, Boumezrag M, Milcamps R, Cohen D. [Visual acuity and ocular diseases in aged residents of nursing homes: study of 219 persons in Orleans]. J Fr Ophtalmol. 1999 May;22(4):431-7. French. PMID 10365330
- [Background] Oeppen J, Vaupel JW. Demography. Broken limits to life expectancy. Science. 2002 May 10;296(5570):1029-31. doi: 10.1126/science.1069675. No abstract available. PMID 12004104
- [Background] Lawrence D, Fedorowicz Z, van Zuuren EJ. Day care versus in-patient surgery for age-related cataract. Cochrane Database Syst Rev. 2015 Nov 2;2015(11):CD004242. doi: 10.1002/14651858.CD004242.pub5. PMID 26524611
- [Background] Laidlaw DA, Harrad RA, Hopper CD, Whitaker A, Donovan JL, Brookes ST, Marsh GW, Peters TJ, Sparrow JM, Frankel SJ. Randomised trial of effectiveness of second eye cataract surgery. Lancet. 1998 Sep 19;352(9132):925-9. doi: 10.1016/s0140-6736(97)12536-3. PMID 9752814
- [Background] Westcott MC, Tuft SJ, Minassian DC. Effect of age on visual outcome following cataract extraction. Br J Ophthalmol. 2000 Dec;84(12):1380-2. doi: 10.1136/bjo.84.12.1380. PMID 11090477